CLINICAL TRIAL: NCT03025269
Title: Effect of Ocrelizumab on Gray Matter Pathology, Leptomeningeal Inflammation and Cognitive Dysfunction in Multiple Sclerosis
Brief Title: Ocrelizumab Effects on Physiological and Cognitive Changes in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, MD, PhD, University at Buffalo
Other Study IDs: STUDY00001202
Record Dates: First submitted 2017-01-16; First posted 2017-01-19 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Relapsing MS patients treated with Ocrelizumab: 30 patients diagnosed with relapsing forms of multiple sclerosis and newly beginning treatment with Ocrelizumab according to neurologists' orders
  Interventions: Drug: Ocrelizumab

INTERVENTIONS:
Drug: Ocrelizumab — This is not a drug intervention study, we are doing an observational study with those who have been prescribed Ocrelizumab by their neurologists during clinical routine appointments

SUMMARY:
This is a Phase IV, prospective, open-label, single-center, observational, longitudinal, single blinded study. The investigators will examine the effects of Ocrelizumab on cognitive, patient reported outcomes (PROs), quality of life (QoL), multiple sclerosis functional composite (MSFC), working status and magnetic resonance imaging (MRI) outcomes across 12 and 24 months.

DETAILED DESCRIPTION:
Grey matter (GM) atrophy develops early in the multiple sclerosis (MS) disease process. Over 2 years, clinically isolated syndrome (CIS) patients developed significant thalamic and cortical volume loss. In our preliminary study, including 50 MS patients, the investigators found that the presence of leptomeningeal (LM) contrast enhancement (CE) was associated with progression of cortical atrophy over 5 years, as measured by the loss of cortical volume, in patients with MS. About 40% of relapsing-remitting MS (RRMS) patients presented with LM CE. MS patients with LM CE showed significantly greater percentage decreases cortical (-3.4% vs. -1.8%, p=0.007) volumes, compared to those without. RRMS patients with LM CE showed significantly greater percentage decrease in cortical (-3.8% vs. -1.9%, p=0.006) volume over the follow-up, compared to those without. No differences in deep GM volume changes were found in relapsing-remitting (RR) and secondary progressive (SP) MS patients with and without LM CE. Three LM CE positive and one LM CE negative RRMS patients developed secondary progressive MS (SPMS) course over the follow-up. More MS subjects with LM CE had disability progression (7, 28%) compared to those without (4, 16%), but this was not significantly different (p=0.306). The median EDSS in MS patient with LM CE increased to 4.0, while decreased to 2.5 in those without. No differences in total number of relapses, annual relapse rate, nor being relapse free were detected in MS patients with and without LM CE over the follow-up. However, in RRMS patients with LM CE, the investigators found that there was a trend for greater increase in absolute change of EDSS (0.9 vs. -0.03, p=0.05).

The proposed study will extend these preliminary findings in a cohort of MS patients, who will be treated with Ocrelizumab and who will be assessed at 12 and 24 months using same MRI hardware and software. The longitudinal serial MRI assessment study design will allow us to examine temporal relationship of LM CE, development of GM pathology, cognitive dysfunction and Ocrelizumab. Based on our preliminary results, the investigators expect that approximately 12 (40%) of MS patients will present with LM CE at baseline in the proposed study.

Substantial evidence shows that Epstein-Barr virus (EBV) infection plays a major role in the risk of developing MS. Mononucleosis and seropositivity of anti-Epstein-Barr nuclear antigen (EBNA) Immunoglobulin G (IgG) along with Vit D deficiency and smoking are risk factors for MS. Serial studies reveal that the risk of developing MS is extremely low among individuals not infected with EBV but increases sharply in the same individuals following EBV infection. EBV-infected B cells were identified in MS brain lesions. Therefore the elimination of the virus from the persistently infected B-cells could potentially inhibit/delay disease progression. Our data show correlation of anti-EBV levels with atrophy (more degeneration) hence an effect on disease chronicity/progression. Besides high Vit D administration studies that showed an effect on decreasing the EBV antibody levels, no other DMT's were able to show a beneficial effect on EBV antibody level, and some treatments increased EBV levels.

EBV viremia occurs in the hematopoietic stem transplantation setting and has been treated successfully with rituximab, an antibody that targets B-lymphocyte antigen (CD20) on B cells in a manner analogous to Ocrelizumab. It has been reported that 92% of patients with EBV viremia responded upon dosing with rituximab and the EBV copies per 100,000 peripheral blood mononuclear cell (PBMC) decreased from 2578 to 71 at Day 15 and 0 by Day 21.

Therefore, our hypothesis is that Ocrelizumab treatment will reduce both B cells and EBV exposure in treated patients leading to benefit on LM inflammation and to less GM atrophy development.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with MS according to McDonald criteria
* Age 18-60
* Relapsing disease course
* Expanded Disability Status Scale (EDSS) ≤5.5
* Disease duration <20 years
* Treatment naive to Ocrelizumab
* Willing and able to comply with the study procedures for the duration of the trial
* Given written informed consent and signed HIPAA Authorization prior to the study
* Normal kidney functioning (creatinine clearance >59)
* None of the exclusion criteria

Exclusion Criteria:

* PI guidelines for contraindications of Ocrelizumab (available after FDA approval)
* Significant cognitive impairment (in the opinion of the investigator) or other significant neurological or medical condition that would compromise adherence and completion of the trial, including major depression and developmental disorders affecting cognition
* Have received treatment within 30 days prior to enrollment with steroids or any other concomitant immunomodulatory therapies
* Have received treatment with Natalizumab within 8 weeks prior to enrollment; this is needed to increase confidence that there are no signs of progressive multifocal leukoencephalopathy (PML) on baseline MRI
* Less than 6 months from the use of immunosuppressant agents (e.g., including but not limited to mitoxantrone, cyclophosphamide, azathioprine, methotrexate, mycophenolate mofetil)
* Have received an investigational drug or experimental procedure within the past 30 days
* Women who are pregnant, lactating, or of childbearing age who do not consent to approved contraceptive use during the study
* Any other factor that, in the opinion of the investigator, would make the subject unsuitable for participation in this study
* Hypersensitivity to trial medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with relapsing multiple sclerosis who are being treated at the Jacobs Neurological Institute (JNI) in Buffalo, NY
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2022-01-08 (Actual); Study Completion 2022-01-08 (Actual)

PRIMARY OUTCOMES:
Absolute cortical atrophy 12 | 12 months
  Absolute change in cortical atrophy between baseline and 12 months
Percent change cortical atrophy 12 | 12 months
  Percent change in cortical atrophy between baseline and 12 months
Absolute cortical atrophy 24 | 24 months
  Absolute change in cortical atrophy between baseline and 24 months
Percent cortical atrophy 24 | 24 months
  Percent change in cortical atrophy between baseline and 24 months
Absolute thalamic atrophy 12 | 12 months
  Absolute change in thalamic atrophy between baseline and 12 months
Percent thalamic atrophy 12 | 12 months
  Percent change in thalamic atrophy between baseline and 12 months
Absolute thalamic atrophy 24 | 24 months
  Absolute change in thalamic atrophy between baseline and 24 months
Percent thalamic atrophy 24 | 24 months
  Percent change in thalamic atrophy between baseline and 24 months
Inflammation foci 12 | 12 months
  Number of leptomeningeal inflammation foci at 12 months
Inflammation foci 24 | 24 months
  Number of leptomeningeal inflammation foci at 24 months

SECONDARY OUTCOMES:
SDMT score 12 | 12 months
  Raw score differences on Symbol Digit Modalities Test score between baseline and 12 months
SDMT 24 | 24 months
  Raw score differences on Symbol Digit Modalities Test score between baseline and 24 months
Memory 12 | 12 months
  Differences in Brief Visuospatial Memory Test Revised between baseline and 12 months
Memory 24 | 24 months
  Differences in Brief Visuospatial Memory Test Revised between baseline and 24 months
Verbal learning 12 | 12 months
  Differences in California Verbal Learning Test Revised between baseline and 12 months
Verbal learning 24 | 24 months
  Differences in California Verbal Learning Test Revised between baseline and 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Jacobs Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No